CLINICAL TRIAL: NCT05463939
Title: Teclistamab US Expanded Access Treatment Protocol for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Teclistamab Expanded Access Treatment Protocol for Relapsed or Refractory Multiple Myeloma Patients
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109154; 64007957MMY4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-07-01; First posted 2022-07-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously (SC).
  Other Names: JNJ-64007957

SUMMARY:
The purpose of this expanded access treatment protocol is to provide patients access to teclistamab prior to market authorization. The program is limited to patients with relapsed or refractory multiple myeloma who have exhausted all treatment options available as local standard of care and who are not eligible for a teclistamab clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Relapsed or Refractory Multiple Myeloma
* Patient exhausted all commercially approved and clinically appropriate (not patient or physician preference) treatment options, and is ineligible for a clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC